CLINICAL TRIAL: NCT03501901
Title: Characteristics of Hospital- and Community-acquired Urinary Tract Infections Caused by ESBL-producing Enterobacteria in a Tertiary-care Hospital
Brief Title: Urinary Tract Infections Caused by ESBL-producing Enterobacteria
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Collaborators: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Soraya Mendoza-Olazarán, Clinical Professor, Universidad Autonoma de Nuevo Leon
Other Study IDs: UR14-004
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Urinary Tract Infections
Keywords: ESBL-producing enterobacteria; hospital- and community-acquired urinary tract infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Biospecimen Retention: Samples Without DNA — Strains of enterobacteria
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Antibiotic susceptibility test

SUMMARY:
The aim of this study was to compare the etiologic agents, the antimicrobial resistance rates, and the risk factors associated with a HA-UTI and CA-UTI among complicated and uncomplicated UTI patients in a tertiary-care hospital in Mexico. This study was performed according to the principles expressed in the Declaration of Helsinki with the approval of the Local Ethics Committee of the School of Medicine of the Universidad Autónoma de Nuevo León (UR14-004). All patients with a UTI and a positive urine culture (> 100,000 UFC/mL) from March to October 2015 were included. The study was carried out at the Hospital Universitario "Dr. José Eleuterio González" hospital, a tertiary-care teaching hospital in Monterrey, Mexico. Identification and susceptibility antibiotic assays were performed to all isolates from positive urine culture.

DETAILED DESCRIPTION:
The aim of this study was to compare the etiologic agents, the antimicrobial resistance rates, and the risk factors associated with a HA-UTI and CA-UTI among complicated and uncomplicated UTI patients in a tertiary-care hospital in Mexico.

This study was performed according to the principles expressed in the Declaration of Helsinki with the approval of the Local Ethics Committee of the School of Medicine of the Universidad Autónoma de Nuevo León (UR14-004).

All patients with a UTI and a positive urine culture (> 100,000 UFC/mL) from March to October 2015 were included. The study was carried out at the Hospital Universitario "Dr. José Eleuterio González" hospital, a tertiary-care teaching hospital in Monterrey, Mexico. This hospital has 500 beds, serves a population of approximately 5 million people, and has an average of 250,000 medical consultations and 22,000 hospitalizations annually.

A UTI was defined as the presence of symptoms related to the urinary tract, pyuria (≥10 leucocytes per high-power field) and a positive urine culture (≥105 CFU/mL) of one uropathogen according to the guidelines of the Infectious Diseases Society of America (IDSA) and the European Association of Urology (EAU). Patients with urine cultures with significative counts of two or more bacterial species were excluded.

Patients' charts were reviewed for clinical and demographic characteristics. The classification of UTIs as either complicated or uncomplicated, and hospital-acquired or community-acquired, was based on the IDSA and EAU criteria. Cases which could not be classified due to insufficient clinical information were excluded.

Urine cultures were performed according to standard protocols. Species identification of all isolates was performed using MALDI-TOF mass spectrometry (Microflex, Bruker Daltonics, Billerica, MA). The drug resistance profile of all E. coli isolates was determined using the broth microdilution method for gentamicin, amoxicillin-clavulanic acid, aztreonam, ceftriaxone, ertapenem, ciprofloxacin, levofloxacin, nitrofurantoin, trimethoprim/sulfamethoxazole, and colistin; except fosfomycin, in which the agar dilution method was used. The results were interpreted according to the Clinical and Laboratory Standards Institute (CLSI) criteria.

Multidrug resistance (MDR) was defined as non-susceptibility to at least one agent in three or more antimicrobial categories. All isolates with resistance to at least one third-generation cephalosporin were evaluated for production of ESBL in E. coli using the double-disc test according to the CLSI.

Categorical variables were expressed as frequencies and percentages. Numerical variables were expressed as a mean and standard deviation. Clinical and demographic characteristics were analyzed using the χ2 test for categorical variables and the t-test (or Mann-Whitney test in the absence of normal distribution) for continuous variables. Statistical significance was set at p <0.05. Statistical analysis was performed with the SPSS software version 20.0 (IBM Corp, Armonk, NY).

ELIGIBILITY:
Inclusion Criteria:

* All patients (> 18 years old) with a UTI and a positive urine culture (> 100,000 UFC/mL) from March to October 2015 were included

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a UTI and a positive urine culture (> 100,000 UFC/mL) from March to October 2015 were included. The study was carried out at the Hospital Universitario "Dr. José Eleuterio González" hospital, a tertiary-care teaching hospital in Monterrey, Mexico. This hospital has 500 beds, serves a population of approximately 5 million people, and has an average of 250,000 medical consultations and 22,000 hospitalizations annually.
Sampling Method: Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Antibiotic resistance | 7 month
  Antibiotic resistance test were perfomed to all Escherichia coli isolates

IPD SHARING:
Plan to Share IPD: Undecided